CLINICAL TRIAL: NCT06165081
Title: The Association Between Post-resuscitation Time Series Management in the Emergency Department and Short-term Outcomes for Out-of-hospital Cardiac Arrest Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202309123RIND
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Resuscitation; Emergency Department; Outcome
Keywords: Out-of-hostpital cardiac arrest; Short-term outcome
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines the impact of emergency department (ED) management on short-term outcomes of nontraumatic adult out-of-hospital cardiac arrest (OHCA) patients. Conducted by a research team at National Taiwan University Hospital and its affiliated hospitals, including branches in Hsinchu and Yunlin, the study spans from January 2016 to August 2023. It focuses on a sequential population of patients, analyzing data like age, gender, medical history, prehospital care details (e.g., witnessed collapse, bystander CPR), and specifics of ED management.

OHCA, with an incidence rate of 50-100 per 100,000 people, presents high mortality and severe complications, leading to significant healthcare expenditures. After resuscitation in the ED, only about one-fifth of patients achieve return of spontaneous circulation (ROSC). The prognosis for these patients remains grim, with a mere 5% experiencing favorable neurological outcomes. Understanding the mechanisms of OHCA, identifying risk factors, effective interventions, and the timing of ED treatments like vasopressors and electrocardiography are crucial.

Patients post-OHCA often undergo a postcardiac arrest syndrome (PCAS), marked by cellular hypoxia and a consequential inflammatory response. Stability of vital signs and rapid ED interventions, including identifying OHCA causes and coordinating with specialists, are vital for short-term recovery. This study aims to determine if ED management and time-related factors from ROSC to various interventions (e.g., ECG, CT scans) affect short-term survival rates, including survival to hospital admission and survival after 1, 3, and 7 days.

By retrospectively analyzing patient data, including Utstein Style prehospital cardiac arrest registry variables and emergency department management details, the study seeks to shed light on the crucial phase of post-resuscitation care. The ultimate goal is to improve survival rates and neurological outcomes in OHCA patients, emphasizing the need for more comprehensive research in this area

DETAILED DESCRIPTION:
The incidence rate of out-of-hospital cardiac arrest (OHCA) is approximately 50 to 100 per 100,000 people. OHCA has a high mortality rate and severe complications that lead to substantial healthcare expenditures. After being resuscitated in the Emergency Department (ED), about one-fifth patients achieve return of spontaneous circulation (ROSC). However, some patients who survive to hospital admission fail to survive. The rate of favorable neurological outcomes is also poor, around 5%. To improve survival rates and neurological outcomes, previous studies focused on understanding the mechanisms of OHCA, identifying risk factors, finding effective interventions, promoting public education, first aid training, and implementing treatments such as targeted temperature management and cardiac catheterization.

OHCA patients experience a postcardiac arrest syndrome (PCAS) between cellular hypoxia and reperfusion, resulting in an inflammatory response in the body. At this stage, patients' vital signs are typically unstable, and emergency department, including initial post-resuscitation care, rapid stabilization of patients, identification of the cause of OHCA and coordination with appropriate specialists, has a significant impact on post-cardiac arrest short-term outcomes. The timing of ED interventions, including the administration of vasopressors, 12-lead electrocardiography, inotropes, and the time-consuming from ROSC to hospital admission, may also influence short-term outcomes. Currently, there is a lack of comprehensive research on whether ED management affects the short-term outcome in OHCA patients. This study highlights the need to collect and analyze information in this regard.

This study is a retrospective study, a series study in our study team, focusing on a sequential population of nontraumatic adult OHCA patients from January 2016 to August 2023 (2016/1/1~2023/8/31) at the National Taiwan University Hospital and its three affiliated hospitals, including branches in Hsinchu and Yunlin. The research variables include basic patient information (age, gender, etc.), past medical history, Utstein Style prehospital cardiac arrest patient registry variables (witnessed collapse, bystander CPR, rhythm, defibrillation, medications, airway management, etc.), emergency department management and time intervals (from ROSC to ECG time, from ROSC to CT time), etc. Primary outcomes include survival to hospital admission, 1-day, 3-day, and 7-day survival rates. This study aims to investigate whether the management of the emergency department and time series factors influences the short-term outcomes in patients following OHCA.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 20 who have experienced cardiac arrest prior to arrival and have been resuscitated to regain spontaneous heartbeat in the emergency department

Exclusion Criteria:

* Traumatic mechanism, Loss of medical record

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research team conducted patient collection at the National Taiwan University (NTU) hospital system, including the NTU Main Hospital, NTU Hsinchu Branch (encompassing the Hsinchu, Zhubei, and Zhudong hospital districts), and NTU Yunlin Branch (covering the Huwei and Douliu hospital districts), totaling three hospitals and six hospital districts. This study aims to collect data on patients who experienced cardiac arrest before arriving at the hospital from January 2016 to August 2023 (1/1/2016 to 8/31/2023)
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained ROSC to hospital admission | 2016/1/1 - 2023/8/31
  The fraction of patient who suffered from OHCA with sustained ROSC to hospital admission (Either ICU or General Ward)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu branch, Hsinchu, Hsinchu City, Taiwan